CLINICAL TRIAL: NCT03255226
Title: A Multicenter, Open-labeled, Dose-defining Trial to Investigate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Tolvaptan in Pediatric Congestive Heart Failure (CHF) Patients With Volume Overload
Brief Title: Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics Study of Tolvaptan in Pediatric Congestive Heart Failure (CHF) Patients With Volume Overload
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-102-00123; JapicCTI-173674 (Other: Japic)
Record Dates: First submitted 2017-08-18; First posted 2017-08-21 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Congestive Heart Failure (CHF) Patients With Volume Overload
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolvaptan (Experimental): Tolvaptan 1% granules or tolvaptan 15 mg tablet with water once daily.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan 1% granules or tolvaptan 15 mg tablet with water once daily.

SUMMARY:
To determine the efficacy, safety, and dose and regimen of tolvaptan in pediatric CHF patients with volume overload

ELIGIBILITY:
Inclusion Criteria:

* Patients with volume overload despite having received any of the following diuretic therapies in whom sufficient effects cannot be expected even if the dose of the diuretics is increased or in whom the investigator or subinvestigator judges that increasing the dose of the diuretics is difficult due to concerns regarding electrolyte abnormalities or other side effects

  * Furosemide (oral administration) ≥0.5 mg/kg/day. Azosemide 30 mg and torasemide 4 mg will be calculated as equivalent to furosemide 20 mg.
  * Hydrochlorothiazide ≥2 mg/kg/day
  * Trichlormethiazide ≥0.05 mg/kg/day
  * Spironolactone ≥ 1 mg/kg/day
* Patients capable of complaining of thirst. Patients unable to complain of thirst due to their young age can also be enrolled in the trial if strict management of fluid intake and excretion is conducted. However, even if such fluid management is possible, the patients in whom the investigator or subinvestigator judges that tolvaptan cannot be safely administered are to be excluded
* Patients who can be hospitalized from at least 3 days before start of tolvaptan administration until 2 days after the final administration.

others

Exclusion Criteria:

* Patients whose volume overload status shows improvement during the screening period or pretreatment observation period
* Patients who are unable to drink fluid (including patients who are unable to sense thirst)
* Patients whose circulatory blood flow is suspected to be decreased
* Patients with an assisted circulation apparatus
* Patients with hypernatremia (serum or blood sodium concentration exceeding 145 mEq/L) others

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kanto Region, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tolvaptan
Started | 60
Completed | 46
Not Completed | 14
Not completed — Adverse Event | 2
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 1
Not completed — Serum or blood sodium increased | 4
Not completed — Serum or blood potassium increased | 4

BASELINE CHARACTERISTICS:
Population: The FAS included 59 of 60 subjects (98.3%) who received the IMP. One subject was excluded from the FAS because the subject received the IMP at least once, and discontinued the trial before the daily urine volume data on Day 1 were obtained.
Arm/Group | Tolvaptan
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.44 (5.03)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 6 months to less than 2 years | 20
  Age group: 2 years to less than 7 years | 16
  Age group: 7 years to less than 15 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 59
Region of Enrollment [Number; unit: participants]
  Japan | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects Whose Was Decreased by 1.7% or More Body Weight From Baseline
Description: The primary endpoint of this trial was the percentage of subjects whose body weight on the day after the third day of treatment with tolvaptan at the evaluation dose (the third day of administration at the evaluation dose) was decreased by 1.7% or more from the weight measured before breakfast (baseline) on the first day of the treatment period (the initial tolvaptan administration day), under the condition that the mean daily urine volume for the 3 days of treatment with tolvaptan at the evaluation dose was higher than the daily urine volume for the pretreatment observation period.
  The percentage of subjects as well as the exact 95% confidence interval (CI) based on binomial distribution were calculated.
Time Frame: Day after Day 3 at evaluation dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 57
percentage of participants | 22.8 [12.7 to 35.8]

2. Secondary Outcome: Change Rate From Baseline in Daily Urine Volume
Description: Daily urine volume was measured for the time interval starting at urination (an instruction to urinate) after breakfast and ending at complete urination immediately before administration on the following day.
  Baseline was 100% and the change rate was calculated like this. Percent change (%) = ([daily urine volume on the Day1, Day2 and Day3 of the tolvaptan at the evaluation dose] - [daily urine volume on baseline] ) / [daily urine volume on baseline] ×100
Time Frame: Baseline, Day1, Day2 and Day3 of administration at evaluation dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of urine volume (mL)
Arm/Group | Tolvaptan
Number analyzed (Participants) | 59
percentage of urine volume (mL)
  Day 1: number analyzed (Participants) | 58
  Day 1 | 53.1 (52.9)
  Day 2: number analyzed (Participants) | 53
  Day 2 | 47.8 (43.3)
  Day 3: number analyzed (Participants) | 46
  Day 3 | 45.8 (29.3)

3. Secondary Outcome: Percent Changes From Baseline in Body Weight (kg)
Description: Percent change from baseline in body weight (kg) on the day after the third day of treatment with tolvaptan at the evaluation dose was evaluated.
  For body weight measured on the day after the third day of administration at the evaluation dose, their percent changes from baseline (before the start of tolvaptan administration on the first day of the treatment period) mean and standard deviation (SD) were calculated.
  Baseline was 100% and the change rate was alculated like this. Percent change (%) = ([body weight on the day after the third day of treatment with tolvaptan at the evaluation dose] - [body weight on baseline] ) / [body weight on baseline] ×100
Time Frame: Day after Day 3 at evaluation dose
Measure: Mean (Standard Deviation); unit: percentage of body weight (kg)
Arm/Group | Tolvaptan
Number analyzed (Participants) | 57
percentage of body weight (kg) | -0.371 (2.470)

4. Secondary Outcome: Improvement Rates of Lower Limb Edema
Description: The improvement rate was defined as the percentage of subjects in whom a symptom was present at baseline and then markedly improved or improved after IMP administration.
  Improvement category is a 4-point scale below:
  * Markedly improved
  * Improved
  * Unchanged
  * Deteriorated
Time Frame: Day after Day 3 at evaluation dose
Population: The FAS included 59 of 60 subjects (98.3%) who received the IMP. One subject was excluded from the FAS because the subject received the IMP at least once, and discontinued the trial before the daily urine volume data on Day 1 were obtained. Number of subjects with lower libm edema at baseline was 35.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 35
percentage of participants | 68.6 [50.7 to 83.1]

5. Secondary Outcome: Improvement Rates of Pulmonary Congestion
Description: as for outcome 4
Time Frame: Day after Day 3 at evaluation dose
Population: The FAS included 59 of 60 subjects (98.3%) who received the IMP. One subject was excluded from the FAS because the subject received the IMP at least once, and discontinued the trial before the daily urine volume data on Day 1 were obtained. Number of subjects with pulmonary conjestion at baseline was 31.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 31
percentage of participants | 51.6 [33.1 to 69.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the start of IMP administration up to 16 days
Description: Subjects who received at least one dose of IMP were included in the safety analysis.
Arm/Group | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 25/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=60)
Cardiac failure chronic (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=60)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiovascular insufficiency (Cardiac disorders) | 1
Erythema of eyelid (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomitng (Gastrointestinal disorders) | 2
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1
Anal erythema (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Thirst (General disorders) | 4
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Blood pressure increased (Investigations) | 1
Blood pressure systolic decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT03255226/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03255226/SAP_001.pdf